CLINICAL TRIAL: NCT04511338
Title: A Randomized, Open Label, Cross-over Feasibility Study for Heparin-free Hemodialysis With the Dialyzer With Endexo™ in End-Stage Renal Disease (ESRD) Subjects
Brief Title: Feasibility Study for Heparin-free Hemodialysis With the Dialyzer With Endexo™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Endexo-002
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-01

CONDITIONS: Chronic Kidney Diseases; Patient Requiring Heparin Free Dialysis Treatments
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sequence AB: circuit A follow by circuit B (Experimental): Circuit (A) includes the dialyzer with Endexo and the CombiSet bloodline Circuit (B) includes dialyzer with Endexo and the Streamline bloodline
  Interventions: Device: Dialyzer with Endexo
- Sequence BA: circuit B follow by circuit A (Experimental): Circuit (B) includes dialyzer with Endexo and the Streamline bloodline Circuit (A) includes the dialyzer with Endexo and the CombiSet bloodline
  Interventions: Device: Dialyzer with Endexo

INTERVENTIONS:
Device: Dialyzer with Endexo — Sequence AB:
  Period 1 Circuit A (Five Visits: 1,2,3,4,5) Period 2 Circuit B (Five Visits: 9,10,11,12,13)
  Sequence BA:
  Period 1 Circuit B (Five Visits: 1,2,3,4,5) Period 2 Circuit A (Five Visits: 9,10,11,12,13)

SUMMARY:
This study will assess the safety and efficacy of heparin free hemodialysis (HD) performed with dialyzers with Endexo in adult end-stage renal disease (ESRD) subjects on thrice-weekly in-center HD.

ELIGIBILITY:
Inclusion Criteria:

1. Must be an adult, defined as having had a 22nd birthday on or before the date of signed informed consent
2. Has been prescribed in center thrice weekly HD for at least 180 days prior to the date of signed informed consent
3. Has been on Conventional HD for at least 30 days prior to the date of signed informed consent. Conventional HD includes: Optiflux dialyzer (F160NR or F180NR), standard of care (SOC) bloodline, Citrasate dialysate, and regularly prescribed heparin dose.
4. Has a prescribed HD treatment duration ≥ 180 minutes (3 hours) and ≤ 270 minutes (4.5 hours) at the time of signed informed consent
5. Has a well-established functional permanent vascular access (AVF, AVG) that can allow a blood flow of at least 250 mL/min
6. Has been on a regularly prescribed heparin dose for HD and has had no change in heparin prescription within 14 days prior to the date of signed informed consent
7. Has the following most recently available laboratory results within 45 days prior to the date of signed informed consent:

   1. Single pool Kt/V (spKt/V) ≥ 1.2
   2. Hemoglobin ≥ 9 g/dL
   3. Platelet count ≥ 100,000/mm3
8. A female of childbearing potential must have a negative serum pregnancy test at the time of screening and agree to use an acceptable method of contraception during the study

Exclusion Criteria:

1. Known allergic reactions to Endexo
2. Known heparin contraindications
3. Hospitalization within 30 days prior to the date of signed informed consent
4. Presence of active malignancy, congestive heart failure New York Heart Association (NYHA) Class III or IV (see Appendix II. A New York Heart Association Functional Classification), or liver cirrhosis
5. Is receiving or has received chemotherapy/radiation therapy/immunotherapy/plasmapheresis therapy within 90 days prior to the date of signed informed consent
6. Is receiving oral or/and intravenous (IV) antibiotics or has used oral or/and IV antibiotics within 14 days prior to the date of signed informed consent
7. Is currently enrolled in or has completed any other investigational product study within 30 days prior to the date of signed informed consent
8. Is receiving anticoagulants including vitamin K antagonists
9. Is receiving a glycoprotein platelet inhibitor
10. Is receiving more than one anti-platelet medication
11. Is receiving systemic heparin therapy for prevention or treatment besides heparin prescribed for dialysis
12. Requiring blood and other labile blood products (for e.g., fresh frozen plasma, platelets) transfusion during HD treatments
13. Has history of clotting or bleeding disorders
14. Has history or current evidence of any condition, therapy, or laboratory abnormality that might interfere with the participant's ability to follow the requirements of the study and participate for the full duration of the study, or is not in the best interest of the subjects to participate, in the opinion of the investigator.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-06-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fresenius Kidney Care Craven County Dialysis Center, New Bern, North Carolina
  - New Bern Dialysis Unit, New Bern, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence AB (Circuit A and Then Circuit B); Sequence BA (Circuit B and Then Circuit A): Circuit (A) includes the dialyzer with Endexo and the CombiSet bloodline
  Dialyzer with Endexo: Sequence AB:
  Period 1 Circuit A (Five Visits: 1,2,3,4,5) Period 2 Circuit B (Five Visits: 9,10,11,12,13)
  Sequence BA:
  Period 1 Circuit B (Five Visits: 1,2,3,4,5) Period 2 Circuit A (Five Visits: 9,10,11,12,13)
Period: Period 1
Arm/Group | Sequence AB (Circuit A and Then Circuit B) | Sequence BA (Circuit B and Then Circuit A)
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0
Period: Washout
Arm/Group | Sequence AB (Circuit A and Then Circuit B) | Sequence BA (Circuit B and Then Circuit A)
Started | 8 (We followed the rules in protocol (brief version in SARP sec. 3.1) to withdraw or move subjects to the next period. Period 1: * Dialyzer with Endexo has grade 4 clotting, subjects is withdrawn from the study * CombiSet with grade 4 clotting only (not the dialyzer): subjects end Period 1, move to Washout, and then Period 2 There was a subject with CombiSet bloodline grade 4 clotting in the 50% heparin reduction HD. The subject was moved to washout period without any heparin free sessions.) | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence AB (Circuit A and Then Circuit B) | Sequence BA (Circuit B and Then Circuit A)
Started | 8 | 8
Completed | 8 | 5
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Sequence AB: Circuit A Following by Circuit B: Circuit (A) includes the dialyzer with Endexo and the CombiSet bloodline
  Dialyzer with Endexo: Sequence AB:
  Period 1 Circuit A (Five Visits: 1,2,3,4,5) Period 2 Circuit B (Five Visits: 9,10,11,12,13)
  Sequence BA:
  Period 1 Circuit B (Five Visits: 1,2,3,4,5) Period 2 Circuit A (Five Visits: 9,10,11,12,13)
- Sequence BA: Circuit B Follow by Circuit A: Circuit (B) includes dialyzer with Endexo and the Streamline bloodline
  Dialyzer with Endexo: Sequence AB:
  Period 1 Circuit A (Five Visits: 1,2,3,4,5) Period 2 Circuit B (Five Visits: 9,10,11,12,13)
  Sequence BA:
  Period 1 Circuit B (Five Visits: 1,2,3,4,5) Period 2 Circuit A (Five Visits: 9,10,11,12,13)
- Total: Total of all reporting groups
Arm/Group | Sequence AB: Circuit A Following by Circuit B | Sequence BA: Circuit B Follow by Circuit A | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (10.16) | 65.0 (6.63) | 64.3 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Number and Percent (%) of Successful Heparin-free HD Sessions for Each Subject in Each Circuit.
Description: Each participant was expected to receive 3 heparin-free HD sessions. The number and percentage of successful HD sessions were derived based on the 3 heparin-free HD sessions for each participant in each circuit.
  A successful HD session must meet all the following criteria:
  1. Absence of complete HD circuit occlusion (Grade 4) rendering dialysis impossible
  2. Absence of the need to replace dialyzers or bloodlines due to clotting
  3. Absence of saline flushes to maintain blood flow through the circuit during the HD session
  4. Absence of any additional heparin beyond what is allowed per study visits
  5. Single pool Kt/V (spKt/V) ≥ 1.2
Time Frame: Approximately 5 weeks, Period 1: two weeks with either Circuit A or Circuit B; Washout: 1 week; Period 2: two weeks with the circuit other than Period 1.
Population: Analysis population, defined as subjects who signed the ICF, met inclusion criteria, did not meet any exclusion criteria, were enrolled, randomized, and had at least one heparin reduction HD treatment.
  Based on the definition of analysis population, there were 15 subjects in Circuit A and 16 subjects in Circuit B.
Measure: Mean (Standard Deviation); unit: number of successful HD sessions
Groups:
- Circuit A: Dialyzer with Endexo + CombiSet bloodline
- Circuit B: Dialyzer with Endexo + Streamline bloodline
Arm/Group | Circuit A | Circuit B
Number analyzed (Participants) | 15 | 16
number of successful HD sessions | 2.4 (1.12) | 2.9 (0.50)

2. Secondary Outcome: The Secondary Endpoints Include Adverse Events .
Description: The number of Serious Adverse Events and Adverse Events during the study periods
Time Frame: two weeks each period (10 weeks per subject: 4 weeks for screening, 2 weeks for Period 1, 1 week for Washout, and 2 weeks for Period 2)
Population: Safety population, defined as subjects who signed the ICF, met inclusion criteria, did not meet any exclusion criteria, were enrolled, and randomized.
  Based on the definition of safety population, there were 16 subjects in Circuit A and 16 subjects in Circuit B.
Measure: Number; unit: events
Arm/Group | Circuit A | Circuit B
Number analyzed (Participants) | 16 | 16
events | 2 | 4

3. Secondary Outcome: The Secondary Endpoints Include Device-related Adverse Events.
Description: All device-related serious adverse events and adverse events occurred during the study periods
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: events
Arm/Group | Circuit A | Circuit B
Number analyzed (Participants) | 16 | 16
events | 0 | 0

4. Other Pre Specified Outcome: Number and Percentage of Dialyzers and Blood Lines for Each Clotting Grade Using the Visual Inspection Clotting Grade Scale
Description: Number and percentage of dialyzers (arterial end cap, venous end cap) and blood lines (CombiSet: Arterial chamber, venous chamber; Streamline: Arterial pod, venous pod, venous chamber) for each clotting grade using the visual inspection clotting grade scale
Time Frame: Approximately 5 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: HD Treatment Duration or Time to Complete Circuit Occlusion (Grade 4)
Description: HD treatment duration or time to complete circuit occlusion (Grade 4). The treatment duration was recorded for each HD session.
Time Frame: Approximately 4.5 hours
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Blood Volume Processed for Heparin Free
Description: Blood volume processed (BVP) for each of 3 heparin free HD sessions (expected). The average of BVPs for each subject was calculated first then the descriptive stat. were derived.
Time Frame: Approximately 4.5 hours for each HD session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Circuit A | Circuit B
Number analyzed (Participants) | 15 | 16
L | 88.33 (7.637) | 92.37 (7.190)

7. Other Pre Specified Outcome: The Volume of Saline Administered Per Subject Per HD Session (Other Than for Circuit Priming or Rinse Back).
Description: The volume of saline administered per subject per HD session (other than for circuit priming or rinse back). The total volume was calculated for each HD session.
Time Frame: Approximately 4.5 hours
Reporting Status: Not Posted

8. Other Pre Specified Outcome: The Time of Saline Administered Per Subject Per HD Session (Other Than for Circuit Priming or Rinse Back).
Description: The time of saline administered per subject per HD session (other than for circuit priming or rinse back) during a HD session.
Time Frame: Approximately 4.5 hours
Reporting Status: Not Posted

9. Other Pre Specified Outcome: The Reason for Saline Administration Per Subject Per HD Session (Other Than for Circuit Priming or Rinse Back).
Description: to determine if a HD was successful. When saline was used for maintaining blood flow or treating clotting, the heparin free HD was not successful.
Time Frame: Approximately 4.5 hours
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Urea Reduction Ratio (URR) for All HD Sessions
Description: to assess the adequacy of each dialysis session
Time Frame: Approximately 5 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: spKt/V for All HD Sessions
Description: to assess the dialysis adequacy of each HD session
Time Frame: 2 weeks for each period
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 2 weeks for each period (10 weeks per subject: 4 weeks for screening period, 2 weeks for Period 1, 1 week for Washout, 2 weeks for Period 2)
Arm/Group | Circuit A | Circuit B
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Circuit A (N=16) | Circuit B (N=16)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT04511338/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT04511338/SAP_001.pdf